CLINICAL TRIAL: NCT04605848
Title: Infrared Thermography Associated With Cutaneous Microcirculation for Detection of Brown-adipose Tissue: Proof of Concept Against PET-CT in Patients Affected by Pheochomocytoma and/or Paraganglioma
Brief Title: Infrared Thermography Associated With Cutaneous Microcirculation for Detection of Brown-adipose Tissue (MICROBAT)
Acronym: MICROBAT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: recruiting problems
Sponsor: University of Avignon (Other)
Collaborators: Centre Hospitalier Henri Duffaut - Avignon (Other); Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UAPV_180620_AVJ
Record Dates: First submitted 2020-10-08; First posted 2020-10-28 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Pheochromocytoma; Paraganglioma
Keywords: pheochomocytoma; brown adipose tissue; infrared thermography; cutaneous microcirculation; PET-CT
MeSH Terms: conditions — Pheochromocytoma; Paraganglioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BAT group (Experimental): Patients will be divided in two groups for statistical analysis:
  * patients with detectable BAT by PET-CT (BAT+)
  * patients with no detectable BAT by PET-CT (BAT-)
  Interventions: Diagnostic Test: Infrared themrography

INTERVENTIONS:
Diagnostic Test: Infrared themrography — measurement of temperature and microcirculation of the skin overlaying BAT depots in the region of FDG-uptake detected by 18F-FDG PET/CT before and after a cold test
  Other Names: Cutaneous microcirculation

SUMMARY:
Patients affected by pheochromocytoma (PHEO) have brown-adipose tissue (BAT) hyperactivation. They perform, in routine settings, a FDG PET-CT scan. The high metabolic activity of BAT and its ability to consume both glucose and fatty acid suggest that it may have potential as a therapeutic target in the treatment of obesity. However, alternative non-invasive techniques to PET-CT BAT detection still need more validation. Accordingly, our aim will be to measure the temperature and microcirculation of the skin overlaying BAT depots in the region of FDG-uptake detected by 18F-FDG PET/CT before and after a cold test in PHEO patients.

DETAILED DESCRIPTION:
Objectives and Methodology:

* To analyse the change in temperature and microcirculation of the skin overlaying BAT depots in the region of FDG-uptake detected by 18F-FDG PET/CT before and after a cold test in PHEO patients.
* To check the decreased temperature and microcirculatory response after a cold test following resection of the tumor

All the patients affected by will benefit from a:

* clinical: treatments
* biological evaluations: glycemia, triglycerides, total cholesterol, HDL-C, LDL-C, plasma epinephrine and norepinephrine, urine catecholamine
* cutaneous microcirculation by means of Laser Speckle Imaging will be recorded at rest and during a cold test in the supra-clavicular region
* cutaneous microcirculation by means of Laser Doppler Flowmetry will be recorded at rest and during a cold test with one probe in the supra-clavicular region and one probe in umbilical region
* skin temperature by means of infrared thermography will be recorded at rest and during a cold test in the supra-clavicular region

Patients who will have surgery will be investigated before and after one year following resection of the tumor.

ELIGIBILITY:
Inclusion Criteria:

* Patients with confirmed pheochromocytoma and/or paraganglioma

Exclusion Criteria:

* pregnant woman
* breastfeeding woman

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2020-07-03 (Actual); Primary Completion 2022-04-29 (Actual); Study Completion 2023-10-20 (Actual)

PRIMARY OUTCOMES:
Skin temperature in supra-clavicular region in basal condition (TSCRbasal) | Day 0
  Skin temperature in supra-clavicular region will be recorded by infrared thermography (FLIR camera) in basal condition
Skin temperature in supra-clavicular region during a cold test (TSCRcold) | Day 0
  Skin temperature in supra-clavicular region will be recorded by infrared thermography (FLIR camera) during a cold test (feet in water at 19°C during 20min)
Baseline difference in skin temperature in supra-clavicular region (diff TSCR) | Day 0
  diff TSCR (day 0) = TSCRcold - TSCRbasal

SECONDARY OUTCOMES:
Cutaneous blood flow in supra-clavicular region in basal condition (PUbasal) | Day 0
  Cutaneous blood flow in supra-clavicular region will be recorded by Laser Speckle Imaging (PeriCam) in basal condition
Cutaneous blood flow in supra-clavicular region during a cold test (PUcold) | Day 0
  Cutaneous blood flow in supra-clavicular region will be recorded by Laser Speckle Imaging (PeriCam) during a cold test (feet in water at 19°C during 20min)
Baseline difference in cutaneous blood flow in supra-clavicular region (∆PU) | Day 0
  diff PU (day0) =PUcold-PUbasal
Volume of Brown Adipose Tissue detected by PET-CT | Day 0
  18FDG PET-CT will be performed and volume will be segmented by PET/CT Viewer..
Activity of Brown Adipose Tissue detected by PET-CT | Day 0
  18FDG PET-CT will be performed and BAT activity (Standardized Uptake Value (SUV) will be segmented by PET/CT Viewer..
Change from baseline difference in skin temperature in supra-clavicular region ( ∆ diffTSCR) at 12 months | Month 12
  ∆ diff TSCR = diff TSCR(month12) - diff TSCR (day0)
Change from baseline difference in cutaneous blood flow in supra-clavicular region ( ∆ diff PU) at 12 months | Month 12
  ∆ diff PU = diff PU (month12) - diff PU (day0)
Volume of Brown Adipose Tissue detected by PET-CT | Month 12
  18FDG PET-CT will be performed and volume will be segmented by PET/CT Viewer..
Activity of Brown Adipose Tissue detected by PET-CT | Month 12
  18FDG PET-CT will be performed and BAT activity (Standardized Uptake Value (SUV) will be segmented by PET/CT Viewer..

CONTACTS AND LOCATIONS:
Overall Officials: Françoise Latil-Plat, Principal Investigator — Centre Hospitalier Henri Duffaut - Avignon
Locations (1):
- Pôle ENDO- Hopital la Conception APHM, Marseille, PACA, France